CLINICAL TRIAL: NCT06730815
Title: Body Image and Physical Activity of Women with Breast Cancer Self-developed Questionnaire-based Follow-up Clinical Trial
Brief Title: Body Image and Physical Activity of Women with Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Other Study IDs: 9533-PTE 2023.
Record Dates: First submitted 2024-12-08; First posted 2024-12-12 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer Female; Physical Inactivity; Quality of Life; Body Image
Keywords: body image after breast cancer; physical activity; life quality
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hungarian women treated for breast cancer

SUMMARY:
The goal of this self-initiated questionnaire-based follow-up clinical trial is to map the body image and physical activity of Hungarian women treated for breast cancer.

The main questions it aims to answer are:

1. How body image changes during different treatments among women treated for breast cancer?
2. How is physical activity among Hungarian women treated for breast cancer?

DETAILED DESCRIPTION:
The aim of our research is to assess the changes in physical activity and body image of women with breast cancer and the impact of these changes on their quality of life using subjective measures, through cross-sectional research and validation of the Body Image After Breast Cancer questionnaire in Hungarian.

ELIGIBILITY:
Inclusion Criteria:

* Adult women diagnosis of breast carcinoma

Exclusion Criteria:

* neuromuscular diseases
* severe congenital musculoskeletal and other disorders
* other surgical procedures within 1 year

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the Department of Oncotherapy in the University of Pécs at the Medical School
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Body Image After Breast Cancer | 1 day
  points, Body Image After Breast Cancer scale contains 53 items in the six main subscales of vulnerability (with twelve items on feelings of the susceptibility of the body to cancer), body stigma (with sixteen items on feeling to hide the body), transparency (with six items on concerns about the obviousness of cancer-related changes to appearance), body limitations (with eight items on feeling about competence and ability), body concerns (with six items on satisfaction about body shape and appearance), and arm concerns (with five items on concerns about arm symptoms and appearance). Items are scored on a five-point Likert scale from "Completely agree" to "Completely disagree" for items 1-23 and from "Never' to "Always" for items 24-53.
  The higher the points, the worse the body image is.
Global Physical Activity Questionnaire | 1 week
  MET-min, Global Physical Activity Questionnaire, GPAQ, 16 questions in 4 topics (assessing work, travel-related and recreational physical activity, and the time of sitting) minimum score: 0 MET-min, maximum score: 15.600 MET-min, the higher the MET-mins, the better the physical activity is.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 | 2 weeks
  Points, the scale has 9 items, 4 point scale (not at all - nearly every day). The sum score 0-27. Scores less than 5 almost always signified the absence of a depressive disorder; scores of 5 to 9 predominantly represented patients with either no depression or subthreshold (i.e., other) depression; scores of 10 to 14 represented a spectrum of patients; and scores of 15 or greater usually indicated major depression. The higher the points, the higher the depression is.
Rosenberg Self-Esteem Scale | 1 day
  Points, 10 items, 0-3 point scales, the sum scale ranges from 0-30. Scores between 15 and 25 are within normal range; scores below 15 suggest low self-esteem. The higher the points, the better the self-esteem is.
Quality of life of cancer patients or survivors (EORTC QLQ-C30) | 1 week
  EORTC QLQ-C30 is a 30-item instrument designed to measure quality of life in all cancer patients. All items scored 1-4 (not at all - to a great extent).
  The higher the points, the worse the quality of life is.
Quality of life of cancer patients or survivors (EORTC QLQ-BR23) | 4 weeks
  EORTC QLQ-BR23 is a 23-item instrument designed to measure quality of life in breast cancer patients. All items scored 1-4 (not at all - to a great extent).
  The higher the points, the worse the quality of life is.
Body Attitudes Test (BAT) | 1 day
  Body Attitudes Test (BAT) has 20 items, all 0-5 points scale (never - always), the sum scale has the minimum of 0, the maximum of 100. The higher the value, the worse the body attitude is.

CONTACTS AND LOCATIONS:
Locations (2):
- Hungary (2):
  - Vörösmarty utca 4., Pécs, Baranya
  - Édesanyák útja 17., Pécs, Baranya

IPD SHARING:
Plan to Share IPD: No